CLINICAL TRIAL: NCT05607615
Title: A Randomized, Placebo-controlled, Double-blind, Parallel-group, 6-Month Study to Evaluate the Safety, Tolerability, and Potential Efficacy of Monthly Trappsol® Cyclo™ Infusions in Patients With Early Alzheimer's Disease
Brief Title: A 6-Month Study to Evaluate the Safety & Potential Efficacy of Trappsol Cyclo in Patients With Early Alzheimer's Disease
Acronym: EAD501
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cyclo Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CTD-TCAD-501
Record Dates: First submitted 2022-10-12; First posted 2022-11-07 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2022-11

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer; Trappsol Cyclo
MeSH Terms: conditions — Alzheimer Disease | interventions — 2-Hydroxypropyl-beta-cyclodextrin

STUDY DESIGN:
Intervention Model Description: This is a randomized, placebo-controlled, double-blind, parallel-group study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple (Participant, Care Provider, Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Intravenous administration over at least 4 hours by IV infusion Trappsol Cyclo either 500 mg/kg or 1000 mg/kg every 4 weeks
  Interventions: Drug: Hydroxypropyl Beta Cyclodextrin
- Placebo (Placebo Comparator): Intravenous administration of 0.5N saline over at least 4 hours every 4 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hydroxypropyl Beta Cyclodextrin — Minimum active dose of 500 mg/kg (equivalent to 18,500 mg/m2) as an intravenous (IV) infusion once every 28 days
  Other Names: Trappsol Cyclo
  Arms: Experimental
Drug: Placebo — 0.5N saline as an intravenous (IV) infusion once every 28 days
  Other Names: 0.5N saline
  Arms: Placebo

SUMMARY:
Approximately 90 patients, aged 50 to 80 years, with a diagnosis of early Alzheimer's disease will take part in this research study. This study will be conducted in the US. There will be 3 treatment groups: 2 Active doses and 1 group will receive placebo completely by chance. Patients, caregiver, Sponsor, nor study staff will know which treatment is assigned. There are 3 periods in this study: Screening to confirm suitability, Treatment to receive study medication, and Follow-up to check overall health post-participation

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, double-blind, parallel-group study that will assess the safety, tolerability, and potential efficacy of Trappsol Cyclo in patients with EAD as defined according to the FDA Guidance for Industry on Early Alzheimer's Disease: Developing Drugs for Treatment. The study will enroll approximately 90 (30 patients/treatment arm) male and female patients aged 50 to 80 years at Screening with characteristic pathophysiologic changes of AD who meet National Institute on Aging-Alzheimer's Association (NIA-AA) criteria for either AD with MCI or mild AD collectively known as EAD (Stages 3 and 4). Enrolled patients must have evidence of progressive cognitive decline in the last year as determined by serial cognitive test scores, if available, or patient or informant/caregiver/study partner (hereafter called caregiver) report as documented by the Investigator

ELIGIBILITY:
Inclusion Criteria:

* MCI due to AD (Stage 3)
* MMSE-2:SV score 20 and 28 at both Screening (V1) and Baseline (V2) with no more than a 3 point change between visits
* Positive PrecivityAD blood test biomarker for AD with high APS (58-100) Locally or centrally read MRI of ARIA

Exclusion Criteria:

* Clinically significant renal disease
* Evidence of a neurodegenerative disease other than AD Severe hypothyroidism
* Abnormally low levels of serum Vitamin B12
* Lacks visual, auditory acuity and/or language abilities adequate to perform cognitive assessments

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-09-23 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Safety assessments to include incidence of Adverse Events and Serious Adverse Events | up to 24 weeks
  Incidence of AEs, SAEs, incidence of abnormal laboratory test results, abnormal ECGs, abnormal physical exams, abnormal vital signs and abnormal hearing assessments assessments

SECONDARY OUTCOMES:
Mean change in total ADAS-Cog-14 score from Baseline | Week 12 and 24
  Memory, Language, and Executive Function
Change in CDR-SB from Baseline | Weeks 12 and 24
  Memory, Orientation, Judgment and Problem Solving, Community Affairs, Home and Hobbies, and Personal Care
Change in MMSE-2:SV total score from Baseline | Weeks 12 and 24
  Orientation, Attention, Memory, Language, and Visual-Spatial Skills
Change in ADCS-CGIC from Baseline | Weeks 12 and 24
  Cognitive, Behavior, and Social and Daily Functioning
Change in ADCS-ADL from Baseline | Weeks 12 and 24
  Basic Activities of Daily Living Items and Instrumental Activities of Daily Living Items

OTHER OUTCOMES:
Change in combined Z-scores from Baseline (V2) to Weeks 12 (V5) and 24 (V8) on ADAS-Cog-14 | At week 12 and week 24
  Memory, Language, and Executive Function
Change in combined Z-scores from Baseline (V2) to Weeks 12 (V5) and 24 (V8) on CDR-SB | At week 12 and week 24
  Memory, Orientation, Judgment and Problem Solving, Community Affairs, Home and Hobbies, and Personal Care
Change in combined Z-scores from Baseline (V2) to Weeks 12 (V5) and 24 (V8) on MMSE-2:SV | At week 12 and week 24
  Orientation, Attention, Memory, Language, and Visual-Spatial Skills
Peak Plasma Concentration (Cmax) | Weeks 4, 8, 12, and 24
  Maximum concentration, determined directly from individual concentration-time data
Time to the Maximum concentration (Tmax) | Weeks 4, 8, 12, and 24
  Time of the maximum concentration, determined directly from individual concentration-time data
Area under the plasma concentration versus time curve (AUC) | Weeks 4, 8, 12, and 24
  Area under the concentration-time curve from time-zero to the time of the last quantifiable concentration

CONTACTS AND LOCATIONS:
Overall Officials: Karen Mullen, MD, Study Director — Cyclo Therapeutics
Locations (5):
- United States (5):
  - Access Research Institute, Brooksville, Florida
  - Charter Research, Winter Park, Florida
  - Tandem/Clincloud, LCC, Marrero, Louisiana
  - Advanced Clinical Institute Inc, Neptune City, New Jersey
  - Wasatch Clinical Research, Salt Lake City, Utah